CLINICAL TRIAL: NCT04102345
Title: Lavender vs Zolpidem: Sleep Quality During Diagnostic Polysomnography
Brief Title: Lavender vs Zolpidem Sleep Quality During Diagnostic PSG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A19-156
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-04

CONDITIONS: Sleep
Keywords: aromatherapy; diagnostic sleep study; zolpidem
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: Non-randomized, pragmatic, clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lavender (Experimental): 1-2 drops of Lavender (essential oil) in approximately 120 ml of distilled water is added to a diffuser 10 minutes before light out. The diffuser runs for approximately 2 hours before automatically being shut off. A low mist option is used on the diffuser.
  Interventions: Other: Lavender Aromatherapy
- Zolpidem (Active Comparator): Pre-prescribed, physician directed use of zolpidem. There is no dose exclusionary criteria for the zolpidem. This study does not have any dose specifications, anyone on zolpidem may be eligible.
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Other: Lavender Aromatherapy — Commercially available lavender essential oil and diffuser.
  Arms: Lavender
Drug: Zolpidem — Physician directed, pre-prescribed. Study team does not prescribe zolpidem.
  Other Names: Ambien
  Arms: Zolpidem

SUMMARY:
In this pragmatic, clinical study the investigators propose that lavender aromatherapy is comparable to Zolpidem (Ambien) in improving the quality of diagnostic sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* In-center diagnostic or split night sleep study (PSG)

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlene E McEvoy, MD, MPH, Principal Investigator — Medical Director, Regions Hospital/HealthPartners Sleep Center
Locations (1):
- Regions Hospital Sleep Center, Maplewood, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lavender | Zolpidem
Started | 26 | 32
Completed | 25 | 32
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lavender | Zolpidem | Total
Number analyzed (Participants) | 25 | 32 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (1639) | 56 (17) | 54.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 22 | 28 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 32 | 57
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a measure of calculated from a person's weight and height.
  kg/m^2 | 33.6 (8.9) | 33.4 (705) | 33.5 (8.1)
Epworth sleepiness scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — ESS measures the general level of daytime sleepiness. ESS consists of eight patient self-reported questions on a 4-point (0-3) scale. The total score ranges from 0-24. A higher score indicates a higher level of daytime sleepiness.
  units on a scale | 8.3 (5) | 7.6 (4.8) | 7.9 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Percentage of total time in bed actually spent in sleep. It is calculated as sum of Stage N1, Stage N2, Stage N3, and REM sleep, divided by the total time in bed and multiplied by 100. A higher percentage is indicative of more efficient sleep.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of time in bed sleeping
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
percentage of time in bed sleeping | 77.6 (15.8) | 76.8 (16.8)

2. Secondary Outcome: Number of Participants With A Successful Polysomnogram (PSG)
Description: A binary outcome (yes/no) based on chart review. The outcome will be inferred from documentation in the chart either in notes or PSG report showing a successful split night or if a diagnosis is made or if a repeat PSG is ordered. Yes is a successful PSG.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
Participants | 24 | 28

3. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: Number of minutes of wakefulness occurring after defined sleep onset. Higher number of minutes indicates a higher WASO or more time awake after onset of sleep.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
minutes | 52.3 (64.2) | 53.7 (60.2)

4. Other Pre Specified Outcome: Total Sleep Time (TST)
Description: Total amount of sleep time scored during the total recording time; includes time from sleep onset to sleep offset and is distributed throughout the sleep time as minutes of Stage N1 sleep, Stage N2 sleep, Stage N3, and rapid eye movement (REM) sleep. A longer total sleep time would be a higher number of minutes.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes of sleep
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
minutes of sleep | 276.9 (134.2) | 254.8 (157.4)

5. Other Pre Specified Outcome: Sleep Onset Latency
Description: Time in minutes from 'lights off' that marks the starting of total recording time to the first epoch scored as sleep. This is how long one takes to fall asleep. A higher number of minutes is indicative of a higher sleep onset latency.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
minutes | 21.8 (13.6) | 15.1 (17.2)

6. Other Pre Specified Outcome: Rapid Eye Movement (REM) Sleep Onset Latency
Description: Rapid eye movement latency is the time in minutes from the sleep onset to the first epoch of REM sleep. This is the time one takes to transition from non-REM to REM sleep. A high number of minutes indicates a longer sleep latency.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
minutes | 145.3 (81.7) | 115.8 (71.7)

7. Other Pre Specified Outcome: Stage 3/4 Sleep Percentage
Description: Percent of time spent in stage N3 sleep. A higher percentage means that one spends more time in stage N3 sleep than the other stages.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of time in stage N3 sleep
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
percentage of time in stage N3 sleep | 17.6 (7.1) | 17.5 (14.3)

8. Other Pre Specified Outcome: Arousal Index
Description: Total number of arousals x 60/TST (min). A higher arousal index indicates a higher number of arousal during the total sleep time.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: arousals
Arm/Group | Lavender | Zolpidem
Number analyzed (Participants) | 25 | 32
arousals | 19.9 (11) | 30.5 (27.9)

ADVERSE EVENTS:
Time Frame: No follow-up. Until completion of PSG, 6-8 hours.
Arm/Group | Lavender | Zolpidem
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/32
Other Adverse Events (participants affected / at risk) | 1/25 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lavender (N=25) | Zolpidem (N=32)
Intolerance to CPAP (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT04102345/Prot_SAP_000.pdf